CLINICAL TRIAL: NCT05149963
Title: The Development of Cognitive Behavioural Therapy (CBT) for Chronic Loneliness in Children and Young People: Protocol for a Single-case Experimental Design
Brief Title: Cognitive Behavioural Therapy (CBT) for Chronic Loneliness in Children and Young People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Holloway University (Other)
Responsible Party: Principal Investigator, Thomas Cawthorne, Trainee Clinical Psychologist, Royal Holloway University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: Royal Holloway Ethics ID: 2498
Record Dates: First submitted 2021-11-13; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Loneliness
Keywords: Loneliness; CBT; Cognitive Behavioural Therapy; Single Case Experimental Design; SCED
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Randomised multiple-baseline Single Case Experimental Design (SCED)
Who Masked: Investigator
Masking Description: The researcher who completes the assessments will be blinded to baseline allocation length
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cognitive Behavioural Therapy (CBT) for Chronic Loneliness (Experimental): Participants will receive an average of 12 50-minute sessions of CBT aiming to reduce their loneliness. The intervention is modular and has been developed for this study. In total there are 10 treatment modules, 1) Assessment, 2) Formulation and Psychoeducation, 3) Challenging Negative Interpersonal Appraisals and Counterproductive Behaviours, 4) Challenging Negative Thoughts and Cognitive Biases, 5) Challenging Self-focussed Attention, Hypervigilance and Camouflaging, 6) Values-based Social-skills Training, 7) Problem Solving, 8) Findings Friends, 9) Managing Emotions and 10) Relapse Prevention. All participants will complete module 1) Assessment and module 2) Formulation and Psychoeducation. They will then work with the clinician to collaboratively develop a treatment plan based on their formulation. The treatment will be comprised of one or more of the intervention modules. All participants will then complete module 10) Relapse Prevention at the end of their treatment.
  Interventions: Other: Cognitive Behavioural Therapy (CBT) for Chronic Loneliness
- Baseline Phase 1 (12 days) (No Intervention): The design of the study is a randomised multiple-baseline single-case experimental design (SCED). Participants will be randomised to one of 4 baseline lengths (12 days, 19 days, 26 days or 33 days). The baseline phase will act as the control condition within and between participants.
- Baseline Phase 2 (19 days) (No Intervention): The design of the study is a randomised multiple-baseline single-case experimental design (SCED). Participants will be randomised to one of 4 baseline lengths (12 days, 19 days, 26 days or 33 days). The baseline phase will act as the control condition within and between participants.
- Baseline Phase 3 (26 days) (No Intervention): The design of the study is a randomised multiple-baseline single-case experimental design (SCED). Participants will be randomised to one of 4 baseline lengths (12 days, 19 days, 26 days or 33 days). The baseline phase will act as the control condition within and between participants.
- Baseline Phase 4 (33 days) (No Intervention): The design of the study is a randomised multiple-baseline single-case experimental design (SCED). Participants will be randomised to one of 4 baseline lengths (12 days, 19 days, 26 days or 33 days). The baseline phase will act as the control condition within and between participants.

INTERVENTIONS:
Other: Cognitive Behavioural Therapy (CBT) for Chronic Loneliness — Participants will receive an average of 12 50-minute sessions of Cognitive Behavioural Therapy (CBT) aiming to reduce their feelings of loneliness
  Arms: Cognitive Behavioural Therapy (CBT) for Chronic Loneliness

SUMMARY:
Loneliness is a significant problem for young people and is associated with a range of physical and mental health difficulties. Meta-analyses have identified that interventions aimed at young people who report loneliness as their primary problem are lacking within the literature. In adults, the most effective interventions for loneliness are those which target the underlying maladaptive social cognitions. Therefore, the investigators have developed a modular Cognitive Behavioural Therapy (CBT) intervention for children and young people aiming to reduce their feelings of loneliness. The aim of this study is to conduct a multiple baseline single-case experimental design (SCED) to assess the efficacy, feasibility and acceptability of this intervention. In total 6-8 11-18-year-olds and their families will be recruited. The design consists of AB+ post-intervention, where A is the baseline phase, B is the intervention phase and then a post-intervention phase. Participants will complete a baseline assessment, before being randomised to one of four different baseline lengths (12 days, 19 days, 26 days or 33 days). Participants will then complete an average of 12 sessions of CBT, with the aim being to reduce their feelings of loneliness over 12 weeks. Participants will then complete a 12-day post-intervention phase. Participant loneliness will be repeatedly assessed throughout the three phases of the intervention using the Three-item Loneliness Scale, which will be the primary outcome. Secondary outcomes will be reliable and clinically meaningful change on the UCLA-LS-3, RCADS and SDQ. Feasibility and participant satisfaction will also be assessed and reported.

DETAILED DESCRIPTION:
The efficacy of CBT for loneliness in children and young people will be evaluated through a randomised multiple-baseline single case experimental design. The design consists of AB+ post-intervention, where A is the baseline phase, B is the intervention phase and then a post-intervention phase. In the SCED approach participants are repeatedly assessed on at least one independent variable, in this case self-reported loneliness on the Three-item Loneliness Scale, across each phase of the intervention. This repeated measurement and within subject replication is then used to test the effects of the intervention for individual participants.

The construction of this SCED trial and the reporting of the results will be in accordance with the Single-Case Reporting Guidelines in Behavioural Intervention (SCRIBE).

Participants will be recruited via advertisements emailed to schools, shared via social media and word of mouth. After consenting, participants and their parents/carers will complete a baseline eligibility assessment. Participants will complete a range of online questionnaires via a secure online platform. Participants will then attend a remote research assessment appointment to determine whether the family meet the eligibility criteria. The researcher completing the baseline and post-intervention assessments will not be involved in the clinical intervention and will be blinded to baseline allocation. After all baseline assessments for the participant group are completed, participants will be discussed within supervision to confirm that the participants meet eligibility criteria. Eligible participants will then be randomised using a random number generator to one of four different baseline lengths (12 days, 19 days, 26 days or 33 days). The decision to have a minimum of 12 observations per phase meets the requirements for guidelines and standards and will allow for sufficient power for Tau-U analysis.

Each of the participating families will then be contacted to inform them of their allocation. Randomisation and contacting of the families will be completed by a third researcher, who is not involved in either the clinical intervention or research assessments. A letter will also be sent to the participants General Practitioner (GP) informing them of the family's participation in the research study. The setting for the entire study will be remote, with both assessments and intervention sessions being conducted remotely a secure video platform.

All participants in the group will begin their baseline phase concurrently. During the baseline phase participants will be asked to complete the Three-Item Loneliness Scale each day via a secure online platform. SMS message reminders will also be sent to the participants and their parent/carers each day.

The baselines phase will be immediately followed by the intervention. Each family will receive (on average) 12 sessions of CBT for loneliness in children and young people. The first 4 sessions will take place bi-weekly, the second 4 sessions weekly and the final 4 sessions fortnightly.

For all participants the first two sessions will be focussed on assessment and then formulation. The final session for all participants will focus on relapse prevention. During the assessment session the participant will be asked to define 3 goal-based outcomes for how participants hope the intervention will reduce their loneliness, which will then guide the treatment process. During the intervention phase the participants will complete routine outcome measures (ROMs) for each session. This will include the Three-Item Loneliness Scale, visual analogue scales (VAS) of mood, anxiety and loneliness and ratings of their goal-based outcomes. The ROMs will be completed via a secure online platform before each session. If participants have not completed the ROMs before their appointment, then participants will be completed with the clinician at the start of the session.

Participants will begin the post-intervention phase immediately after the final session of their intervention. During the post-intervention phase participants will be asked to complete the primary outcome measure, Three-Item Loneliness Scale each day for 12 days. Participants will then complete their post-intervention assessment with the second researcher. Before the assessment participants will be asked to re-complete the baseline questionnaires in addition to the parent and child-report versions of the Experience of Service Questionnaire and a questionnaire asking whether COVID-19 or any other events have affected their loneliness during the intervention period. A letter will be sent to the participants General Practitioner (GP) informing them of their participation in the research study has finished.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged 11-18
2. Score more than 42 on the UCLA-LS-3 (Russel, 1996), which is more than one standard deviation above the mean in a large community adolescent sample (Shevlin, 2015).
3. Have a parent/carer who is willing to take part in the study.
4. Report loneliness as their primary difficulty (i.e., they are able to identify relevant goal-based outcomes and their current difficulties are not attributable to a significant mental health problem).

Exclusion Criteria:

1. Currently receiving psychological therapy.
2. Started taking antidepressant in the last 8 weeks.
3. Eligibility assessment indicates a severe mental health problem not considered suitable for the trial intervention due to the clinical need for immediate intervention, e.g., active suicidality and psychosis.
4. Refusal for therapy sessions to be video recorded.
5. Having an intellectual disability at a level whereby they cannot access the intervention
6. Do not have access to a laptop or smartphone which they can use for video calls.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Estimated)
Dates: Start 2020-05-27 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in scores on the Three Item Loneliness Scale (Klein et al., 2021) across the baseline, intervention and post-intervention phases. | This study is a single-case experimental design. Participants will complete the measure daily during the baseline phase, each session during the intervention phase, and daily during the post-intervention.
  Self-reported child loneliness. The scale is a brief three-item measure with possible scores ranging from 0-12, with higher scores indicating higher levels of loneliness.

SECONDARY OUTCOMES:
UCLA-Loneliness Scale-3 (Russell, 1996) | Completed at baseline and post-intervention assessments at study completion an average of 16 weeks later.
  Self-reported child loneliness. Scores range from 0-60, with higher scores indicating higher levels of loneliness.
The Strengths and Difficulties Questionnaires (SDQ) (Goodman, 2001) | Completed at baseline and post-intervention assessments at study completion an average of 16 weeks later.
  Parent and self-reported child mental wellbeing. Scores range from 0-40, with higher scores indicating higher levels of difficulty.
The Revised Child Anxiety and Depression Scale (RCADS) (Chorpita et al., 2000) | Completed at baseline and post-intervention assessments at study completion an average of 16 weeks later.
  Parent and self-reported child anxiety and depression. Raw scores are converted into age and gender specific T-scores, with higher scores indicating higher levels of difficulty.

OTHER OUTCOMES:
Goal based outcomes (Law & Jacob, 2013) | This will be completed each intervention session over an average of 12 weeks.
  During their first intervention session young people will be asked to identify 3 intervention goals relating to their loneliness. They will be asked to rate on a 1-10 scale where they are in terms of achieving this goal; with 1 being "the furthest I could ever be from achieving this goal" and 10 "I have achieved this goal".
Visual analogue scales (VAS; see Wewers & Lowe, 1990 for review) | This will be completed each intervention session over an average of 12 weeks.
  For each session young people will be asked to rate their current mood, anxiety and loneliness on a 1-10 scale, where 10 is the worst.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Holloway, University of London, Egham, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymised data will be made available to other researchers on request and the research ethics committee will be informed.
Supporting Information: Study Protocol
Time Frame: We are currently in the process of publishing the study protocol. It will be publish Open Access and available for free.

REFERENCES:
- [Background] Klein, E. M., Zenger, M., Tibubos, A. N., Ernst, M., Reiner, I., Schmalbach, B., ... & Beutel, M. E. (2021). Loneliness and its relation to mental health in the general population: Validation and norm values of a brief measure. Journal of Affective Disorders Reports, 4, 100120.
- [Background] Chorpita BF, Moffitt CE, Gray J. Psychometric properties of the Revised Child Anxiety and Depression Scale in a clinical sample. Behav Res Ther. 2005 Mar;43(3):309-22. doi: 10.1016/j.brat.2004.02.004. PMID 15680928
- [Background] Goodman R. Psychometric properties of the strengths and difficulties questionnaire. J Am Acad Child Adolesc Psychiatry. 2001 Nov;40(11):1337-45. doi: 10.1097/00004583-200111000-00015. PMID 11699809
- [Background] Russell DW. UCLA Loneliness Scale (Version 3): reliability, validity, and factor structure. J Pers Assess. 1996 Feb;66(1):20-40. doi: 10.1207/s15327752jpa6601_2. PMID 8576833
- [Background] Wewers ME, Lowe NK. A critical review of visual analogue scales in the measurement of clinical phenomena. Res Nurs Health. 1990 Aug;13(4):227-36. doi: 10.1002/nur.4770130405. PMID 2197679
- [Background] Law, D., & Jacob, J. (2013). Goals and goal based outcomes (GBOs). London: CAMHS Press.
- [Background] Kazdin AE. Single-case experimental designs. Evaluating interventions in research and clinical practice. Behav Res Ther. 2019 Jun;117:3-17. doi: 10.1016/j.brat.2018.11.015. Epub 2018 Dec 2. PMID 30527785
- [Background] Tate RL, Perdices M, Rosenkoetter U, Shadish W, Vohra S, Barlow DH, Horner R, Kazdin A, Kratochwill T, McDonald S, Sampson M, Shamseer L, Togher L, Albin R, Backman C, Douglas J, Evans JJ, Gast D, Manolov R, Mitchell G, Nickels L, Nikles J, Ownsworth T, Rose M, Schmid CH, Wilson B. The Single-Case Reporting Guideline In BEhavioural Interventions (SCRIBE) 2016 Statement. Phys Ther. 2016 Jul;96(7):e1-e10. doi: 10.2522/ptj.2016.96.7.e1. PMID 27371692
- [Background] Parker RI, Vannest KJ, Davis JL, Sauber SB. Combining nonoverlap and trend for single-case research: Tau-U. Behav Ther. 2011 Jun;42(2):284-99. doi: 10.1016/j.beth.2010.08.006. Epub 2011 Feb 3. PMID 21496513
- [Derived] Cawthorne T, Kall A, Bennett S, Andersson G, Shafran R. The development of Cognitive Behavioural Therapy (CBT) for chronic loneliness in children and young people: Protocol for a single-case experimental design. PLoS One. 2022 Dec 9;17(12):e0278746. doi: 10.1371/journal.pone.0278746. eCollection 2022. PMID 36490292